CLINICAL TRIAL: NCT06580379
Title: Spine Surgery Video Observation Study. The Creation of a Benchmark Video (RGB-Depth) Dataset to Investigate the Feasibility of Developing a Markerless Tracking System for Spine Surgery.
Acronym: SPIVOS
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 168041
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Spine Fusion; Spine Injury; Spine Degeneration; Navigation, Spatial
Keywords: Imaging; Depth Imaging; Spine Surgery; Intraoperative Registration
MeSH Terms: conditions — Spinal Injuries; Spatial Navigation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spine Surgery Patients: non-vulnerable adults undergoing spine surgery, with a posterior approach
  Interventions: Procedure: Spine surgery

INTERVENTIONS:
Procedure: Spine surgery — Spine surgery, such as fusion requiring the need for precise intraoperative registration and navigation

SUMMARY:
The primary study objective is to build a video dataset, consisting of both colour and depth information, of spine surgery that includes both 'open' and 'minimally invasive' (MIS) surgeries. Using accompanying preoperative CT scans of the patient's spine, we aim to develop a markerless tracking system for spine surgery, which the collected dataset will be used to both train, and then benchmark against.

ELIGIBILITY:
Inclusion Criteria:

* Candidate surgeries include all spine surgeries taking a posterior approach. This includes both 'open' and 'minimally invasive' surgeries, provided some portion of vertebrae bone is exposed.

Exclusion Criteria:

* Candidate surgeries will be excluded if the patient is under the age of 18 or the clinical lead feels the patient lacks capacity to consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult spine surgery candidates treated within the Imperial College Healthcare NHS Trust , with the capacity to consent (non-vulnerable)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of Data Collection completed | 3 years (initial recording duration)
  Success in recording 25 RGB-D videos of spine surgeries along with corresponding CT scans
Number of Data points collected containing a variety of exposed spine anatomy | 3 years (initial recording duration)
  Collected samples should contain a wide variety of exposed vertebrae, including cervical, thoracic and lumbar vertebrae
Patient diversity in Ethnicity | 3 years (initial recording duration)
  Patients undergoing surgery should be diverse in terms of ethnicity, diversity being the % of patients who are not 'white british'
Patient diversity in Age | 3 years (initial recording duration)
  Patients undergoing surgery should be diverse in terms of age, diversity being captured by range and standard deviation measures

SECONDARY OUTCOMES:
Usefulness for training navigation system | 4 years (initial recording duration + 1)
  Outcome is to leverage the recordings to train a markerless tracking system that will intraoperatively track the pose and location of the spine within the surgical site. The trained system will be benchmarked against a test subset of the collected videos. The success of the trained system will be determined by its accuracy in automatically tracking the pose of vertebrae features within the test subset videos, against the labelled pose indicated in the video by the operating surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Russo, MD, Principal Investigator — Imperial College Healthcare Trust

IPD SHARING:
Plan to Share IPD: No
There is no plan as of yet to share IPD